CLINICAL TRIAL: NCT07372924
Title: A Phase II, Multicenter, Randomized, Single-Blind, Dose Exploration, Positive Comparator Study to Evaluate the Efficacy and Safety of Tegileridine Fumarate Lnjection for Prolonged Mechanical Ventilation Abirritation in the Intensive Care Unit (ICU)
Brief Title: A Trial of Tegileridine Fumarate Lnjection for Prolonged Mechanical Ventilation Abirritation in the Intensive Care Unit (ICU)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8554-205
Record Dates: First submitted 2026-01-04; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Abirritation in the ICU
MeSH Terms: interventions — Remifentanil; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: Tegileridine Fumarate lnjection (Experimental)
  Interventions: Drug: Tegileridine Fumarate lnjection
- Treatment group B: Tegileridine Fumarate lnjection (Experimental)
  Interventions: Drug: Tegileridine Fumarate lnjection
- Treatment group C: Remifentanil Hydrochloride for Injection (Active Comparator)
  Interventions: Drug: Remifentanil Hydrochloride for Injection

INTERVENTIONS:
Drug: Tegileridine Fumarate lnjection — Tegileridine Fumarate lnjection; low dose
  Arms: Treatment group A: Tegileridine Fumarate lnjection
Drug: Tegileridine Fumarate lnjection — Tegileridine Fumarate lnjection; high dose
  Arms: Treatment group B: Tegileridine Fumarate lnjection
Drug: Remifentanil Hydrochloride for Injection — Remifentanil Hydrochloride for Injection
  Arms: Treatment group C: Remifentanil Hydrochloride for Injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Tegileridine Fumarate lnjection for prolonged abirritation(48h to 72h) during mechanical ventilation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their guardians are able to provide a written informed consent
2. Subjects have been treated with endotracheal intubation and mechanical ventilation ≤24h, and then prolonged mechanical ventilation ≥48h in the next
3. Age ≥ 18 and ≤ 85 years, Male or female
4. Body mass index (BMI) > 18 and < 30 kg/m2
5. Use of highly effective contraception for a specified period if applicable

Exclusion Criteria:

1. Those who are known or suspected to be allergic or contraindicated to various components of the experimental drugs involved in the research institute
2. With an expected survival time of less than 48 hours
3. unable to undergo CPOT and RASS assessments due to various reasons, such as a history of psychiatric disorders, neurological disorders, neurological dysfunction, and consciousness disorders, as well as blindness, deafness, or aphasia
4. Myasthenia gravis, bronchial asthma attack, acute intestinal obstruction, abdominal compartment syndrome
5. Multiple organ failure
6. Malignant tumor Subjects who received radiotherapy, chemotherapy, targeted therapy, and immunotherapy within the first month of randomization
7. Chronic pain requires long-term use of analgesics
8. Severe liver dysfunction
9. Severe renal dysfunction
10. Severe renal dysfunction
11. Need to receive deep sedation or use neuromuscular blocking drugs
12. Surgery or tracheotomy may be required during the study administration period
13. Used monoamine oxidase inhibitors within the two weeks randomization
14. History of drug abuse, drug use, alcohol abuse, and long-term use of psychotropic drugs within 2 years prior to the start of the screening period
15. QTc abnormality during screening period
16. Positive result for infectious disease
17. Positive screening for drug abuse
18. Pregnant or nursing women;
19. Subjects who has Participated in any other clinical trials within the first 3 months of randomization
20. Other conditions deemed unsuitable to be included.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of abirritation success, abirritation success is defined as the percentage of time maintaining target abirritation in the entire drug administering time ≥ 70%. | within 3 days after administration of research drug

SECONDARY OUTCOMES:
Percentage of time maintaining target abirritation in the entire drug administering time. | within 3 days after administration of research drug
Percentage of subjects receiving rescue analgesic drug | within 3 days after administration of research drug
The total dosage of rescue analgesic drug | within 3 days after administration of research drug
Receiving the total dosage of sedation | within 3 days after administration of research drug
Nursing Scores | within 3 days after discontinuation of research drug
  The investigator will conduct an overall nursing assessment of the subject during the safety follow-up period, and the sum of each score will be calculated : (1) Overall Assessment of Adaptability to Sedation and the Intensive Care Environment, Very Easy=1, Easy =2, Fair =3, Difficult=4; (2) Overall Assessment of Adaptability to Endotracheal Intubation/Ventilation, Good=1, Fair =2,Poor=3; (3) Overall Assessment of Ease of Communication with the Patient, Very Easy=1, Easy =2, Fair =3, Difficult=4, Impossible=5; (4) Overall Assessment of Ease of Patient Care, Good=1, Fair =2,Poor=3.
Mechanical ventilation time. | From research drug administration to actual extubation , up to 72 hours
Extubation time | From discontinuation of research drug to actual extubation , up to 72 hours

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Hubei, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided